CLINICAL TRIAL: NCT02946359
Title: Crizotinib Combined With Bevacizumab as First-line Therapy in Metastatic Lung Adenocarcinoma Cancer With ALK Translocation or MET Amplification or ROS1 Translocation (CAMAR)
Brief Title: A+C in Metastatic Lung Adenocarcinoma Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, yihu, Director of oncology department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMAR01
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Lung Adenocarcinoma Metastatic
MeSH Terms: interventions — Crizotinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patients with ALK translocation (Experimental): Treatment-naive lung adenocarcinoma cancer patients with ALK translocation with locally advanced or metastatic lung adenocarcinoma cancer and with at least one measurable tumor lesion will be considered eligible for the trial and they will receive crizotinib 250 mg BID p.o combined with bevacizomab 7.5mg/kg every three weeks until disease progression, unacceptable toxicity or patient refusal
  Interventions: Drug: Crizotinib, bevacizumab
- Patients with ROS1 translocation (Experimental): Treatment-naive lung adenocarcinoma cancer patients with ROS1 translocation with locally advanced or metastatic lung adenocarcinoma cancer and with at least one measurable tumor lesion will be considered eligible for the trial and they will receive crizotinib 250 mg BID p.o combined with bevacizomab 7.5mg/kg every three weeks until disease progression, unacceptable toxicity or patient refusal
  Interventions: Drug: Crizotinib, bevacizumab
- Patients with MET amplification (Experimental): Treatment-naive lung adenocarcinoma cancer patients with MET amplication with locally advanced or metastatic lung adenocarcinoma cancer and with at least one measurable tumor lesion will be considered eligible for the trial and they will receive crizotinib 250 mg BID p.o combined with bevacizomab 7.5mg/kg every three weeks until disease progression, unacceptable toxicity or patient refusal
  Interventions: Drug: Crizotinib, bevacizumab

INTERVENTIONS:
Drug: Crizotinib, bevacizumab — Eligible patients with ALK translocation or ROS1 translocation or MET amplification will be treated with Crizotinib at the standard dose of 250 mg BID and bevacizumab at the dose of 7.5mg/kg every three weeks. The dose of crizotinib and bevacizumab may be adjusted depending on the type and severity of toxicity encountered
  Other Names: XALKORI,AVASTIN

SUMMARY:
This is a phase II, prospective, single arm, non comparative study with crizotinib combined with bevacizumab in treatment-naive lung adenocarcinoma cancer patients with ALK translocation or ROS1 translocation or MET amplification

DETAILED DESCRIPTION:
This is a phase II, prospective, single arm, non comparative study with crizotinib combined with bevacizumab in treatment-naive lung adenocarcinoma cancer patients with ALK translocation or ROS1 translocation or MET amplification. Patients with locally advanced or metastatic NSCLC(Stage ⅢB/ⅢC/Ⅳ) with at least one measurable tumor lesion will be considered eligible for the trial. All potentially eligible patients will be evaluated for ALK、MET and ROS1 by FISH or IHC or NGS to detect MET amplification or ALK translocation or ROS1 translocation After evaluation of inclusion and exclusion criteria, and after signature of informed consent form, all MET amplified or ALK translocation or ROS1 translocated eligible patients will receive crizotinib 250 mg BID p.o and bevacizumab 7.5mg/kg every three weeks until disease progression, unacceptable toxicity or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of lung adenocarcinoma cancer
* Availability of tumor tissue for ROS1, ALK, MET analyses
* EGFR was wild type, positive for ROS1 translocation or ALK translocation or MET amplification
* At least one radiological measurable disease according to RECIST criteria (Response Evaluation Criteria in Solid Tumors )
* Patient didn't received any therapy for lung cancer before except surgery or radiotherapy, or the adjuvant chemotherapy had stopped for more than 12 months
* Performance status 0-2 (ECOG)
* Patient compliance to trial procedures
* age ≥ 18 years
* Written informed consent
* Adequate BM function (ANC ≥ 1.5x109/L, Platelets ≥ 100x109/L, HgB > 9g/dl)
* Adequate liver function (bilirubin <G2, transaminases no more than 3xULN/<5xULN in present of liver metastases).
* Normal level of alkaline phosphatase and creatinine.
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of approved contraceptive method [intrauterine contraceptive device (IUD), birth control pills, or barrier device] during and for ninety(90) days after end of treatment.

Exclusion Criteria:

* Patients with EGFR mutation
* No tumor tissue available or patient negative for ALK translocation or ROS1 translocation or MET amplification
* Absence of any measurable lesion
* Prior therapy with bevacizumab or ipilimumab
* Symptomatic brain metastases
* Previous radiotherapy on the target lesion(s). If all sites were included in radiotherapy fields patient is eligible only if there is evidence of progressive disease after completion of radiotherapy.
* Diagnosis of any other malignancy during the last 5 years, except for in situ carcinoma of cervix uteri and squamous cell carcinoma of the skin
* Pregnancy or lactating
* Other serious illness or medical condition potentially interfering with the study
* Significant known vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure or significant traumatic injury within 28 days prior to study enrollment
* Serious, non-healing wound, ulcer or bone fracture
* Proteinuria at screening
* Known hypersensitivity to any component of bevacizumab
* History of hemoptysis within 3 months prior to study enrollment
* Current, ongoing treatment with full-dose warfarin or its equivalent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-10 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months
Response rate in patients with ALK translocation or ROS1 translocation or MET amplification | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months
Toxicity analysis: Incidence of Grade 3-4 Grade Toxicity graded according to National Cancer | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 months
  Incidence of Grade 3-4 Grade Toxicity graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - PLA general hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided